CLINICAL TRIAL: NCT04586452
Title: CCR2 Targeted Molecular Imaging and Treatment of Abdominal Aortic Aneurysms
Brief Title: NIH CCR2 AAA Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202008190
Record Dates: First submitted 2020-09-29; First posted 2020-10-14 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Abdominal Aortic Aneurysm (AAA); No Abdominal Aortic Aneurysm (Non-AAA)
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Receptors, CCR2

STUDY DESIGN:
Intervention Model Description: There are two (2) groups in the study.
  AAA Group: 40 (20 men; 20 women) participants who will have a PET/CT imaging study performed and a subset of 20 participants who will have an additional PET/CT imaging study performed.
  Non-AAA Group: 10 without AAA (5 men; 5 women), above the age of 40, with or without active tobacco use
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- AAA Group (Aim 3A) (Experimental): 40 (20 men; 20 women) participants with a diagnosis of AAA (above 40 years) will undergo a PET/CT scan prior to their scheduled surgical repair of their condition. The radiotracer, 64Cu-DOTA-ECL1i, will be injected to detect CCR2+ inflammatory cells. A dosage range of 8-10 mCi (296-370 MBq) is planned for 64Cu-DOTA-ECL1i. A PET-certified medical professional will draw and administer the 64Cu-DOTA-ECL1i tracer. The dosage will be assayed in a dose calibrator before and after the administration.
  Interventions: Diagnostic Test: AAA Group (Aim 3A)
- Non-AAA Group (Experimental): 10 (5 men; 5 women) participants will have a documented absence of AAA by screening ultrasound that was previously obtained as part of standard of care. A dosage range of 8-10 mCi (296-370 MBq) is planned for 64Cu-DOTA-ECL1i. A PET-certified medical professional will draw and administer the 64Cu-DOTA-ECL1i tracer. The dosage will be assayed in a dose calibrator before and after the administration.
  Interventions: Diagnostic Test: Non-AAA Group
- Ex Vivo Human AAA Specimens (Aim 2A) (Other): Tissue samples obtained from an existing tissue bank as well as discarded tissue obtained from participants in this study will be examined to assess the sensitivity and specificity of 64Cu-DOTA-ECL1i binding to ex vivo to human AAA specimens.
  Interventions: Other: Ex Vivo Human AAA Specimens (Aim 2A)
- Radiotracer and CCR2 (Aim 2B) (Other): Tissue samples obtained from an existing tissue bank as well as discarded tissue obtained from participants in this study will be examined to better understand the relationship between the levels of CCR2+ inflammatory cells and the inflammatory and clinical status of AAA, to gain insight into the importance of proinflammatory monocytes/macrophages in the development of AAA disease at the time of elective AAA repair.
  Interventions: Other: Relationship between radiotracer and CCR2 (Aim 2B)
- AAA Group (Aim 3B-Reproducibility) (Experimental): 20 (10 men; 10 women) will receive a second PET/CT imaging study performed 10-14 days after the first PET/CT in order to determine the ability to reproduce the uptake results. A dosage range of 8-10 mCi (296-370 MBq) is planned for 64Cu-DOTA-ECL1i. A PET-certified medical professional will draw and administer the 64Cu-DOTA-ECL1i tracer. The dosage will be assayed in a dose calibrator before and after the administration.
  Interventions: Diagnostic Test: AAA Group (Aim 3B-Reproducibility)

INTERVENTIONS:
Diagnostic Test: AAA Group (Aim 3A) — The primary goal is to relate preoperative 64Cu-DOTA-ECL1i AAA uptake with CCR2+ cell activity in AAA tissue collected at the time of open repair. We will image AAA patients pre-operatively and collect tissue at the time of open repair in an attempt to demonstrate ex-vivo tissue corroboration of our imaging findings (n=20, 10 women and 10 men).
  Participants with AAA will undergo routine clinical evaluation including ultrasound, CT scan and scheduling of open surgical repair. We will record age and tobacco use. If a renal function blood test has not been performed within the past 90 days, we will draw ~2 teaspoons of blood for a creatinine test. A contrast dye will be used for the CT portion of the PET-CT scan. Those having open surgery, their PET/CT imaging will be within 7-14 of the surgery and if available, collection of discarded aortic tissue at the time of surgery.
  Arms: AAA Group (Aim 3A)
Diagnostic Test: Non-AAA Group — We will determine the retention of 64Cu-DOTA-ECL1i in abdominal aorta of non-AAA volunteers (n=10, 5 women and 5 men). This group of participants will have a documented absence of AAA by screening ultrasound that was previously obtained as part of standard care. Both men and women, above the age of 40, with or without active tobacco use will be considered for participation.
  Arms: Non-AAA Group
Other: Ex Vivo Human AAA Specimens (Aim 2A) — The primary objective of this sub-aim is to assess the sensitivity and specificity of 64Cu-DOTA-ECL1i binding to ex vivo to human AAA specimens from the Washington University Vascular Surgery Biobank (VS-BB). We will first perform a histopathological evaluation of human AAA specimens (n=75, including samples from this study) and categorize them based on clinical status (e.g, diameter) and degree of inflammation. We will consider healthy, nonatherosclerotic aorta (n=25) as negative controls, and non-aneurysmal aortas (n=25) from patients that have undergone surgery for aortoiliac occlusive disease as positive controls.
  Arms: Ex Vivo Human AAA Specimens (Aim 2A)
Other: Relationship between radiotracer and CCR2 (Aim 2B) — The objective of this sub-aim is to better understand the relationship between the levels of CCR2+ inflammatory cells and the inflammatory and clinical status of AAA, to gain insight into the importance of proinflammatory monocytes/macrophages in the development of AAA disease at the time of elective AAA repair. We will correlate the level of MMP expression and activity, as well as cytokine profiles, of each specimen, with the associated histopathological features. The relationship between 64Cu-DOTA-ECL1i binding and CCR2 expression in tissues with different degrees of disease severity will be evaluated using Pearson or Spearman correlation coefficients. This will allow us to speculate as to how tracer uptake will perform in vivo and what that uptake represents in regard to disease severity.
  Arms: Radiotracer and CCR2 (Aim 2B)
Diagnostic Test: AAA Group (Aim 3B-Reproducibility) — We will demonstrate consistent 64Cu-DOTAECL1i uptake by performing repeated imaging studies in a separate group of non-surgical AAA patients (n=20, 10 women and 10 men). Completion of this sub-aim will provide support for the use of 64Cu-DOTA-ECL1i PET for evaluating AAA disease in a reliable fashion. These participants will have another PET/CT imaging study performed 10-14 days after the first PET/CT in order to determine the ability to reproduce the uptake results of Cu-64-DOTA-ECL1i. The physician will assess the participant's willingness and eligibility to have a second PET/CT scan.
  Other Names: Reproducibility
  Arms: AAA Group (Aim 3B-Reproducibility)

SUMMARY:
Abdominal aortic aneurysm (AAA) is a degenerative vascular disease, which is typically asymptomatic until rupture, resulting in high mortality. AAAs are more prevalent in men over age 65, though rupture is disproportionately higher in women. Due to nonlinear and unpredictable aortic dilatation, it is challenging to predict the AAA rupture using clinical diagnostics based on morphology. No medical therapy is used clinically to treat AAA, and there is an unmet need for clinically translatable, molecular biomarkers of AAA disease activity for surveillance and patient-specific management. The goal of this proposal is to develop a new approach for the diagnosis and targeted therapy of AAA.

DETAILED DESCRIPTION:
This project addresses the absence of a reliable diagnostic modality and medical therapy to prevent abdominal aortic aneurysm (AAA) growth and rupture in patients, leading to high mortality in those over the age of 65 years old. Due to the pathogenic role of the monocyte chemoattractant protein-1 / C-C chemokine receptor type 2 (MCP-1/CCR2) axis in AAA, we propose to study the ability of 64Cu-DOTA-ECL1i PET/CT to predict the murine AAA rupture and serve as a companion diagnostic to assess CCR2 molecular therapy of murine AAA. We will perform the first-in-patient evaluation of 64Cu-DOTA-ECL1i PET/CT to image and detect AAA inflammation in a preoperative setting and acquire key biological information from AAA specimens collected at the time of open AAA repair, in order to assess the potential of 64Cu-DOTA-ECL1i PET in the management of AAA patients.

Preclinical and clinical research demonstrated that monocyte chemotactic protein-1/ chemokine (C-C motif) receptor 2 (MCP-1/CCR2) plays an important role in the pathogenesis of AAAs. This axis specifically promotes AAA formation and development by mediating the recruitment of circulating LY6Chigh monocytes and infiltration of macrophages, which leads to the degradation of elastic and collagen. In AAA mouse models, the genetic depletion or specific inhibition of CCR2 significantly decreased the production of matrix metalloproteinases (MMPs) and formation of aneurysms, suggesting the potential of CCR2 as a biomarker for AAA imaging and pre-screening for targeted intervention.

We have developed a specific CCR2 binding radiotracer, 64Cu-DOTA-ECL1i, for targeted imaging of CCR2 positive pro-inflammatory monocytes/macrophages, in multiple animal inflammatory models using positron emission tomography (PET). This investigational PET tracer is being used under Exploratory IND 137620 for research imaging studies in human subjects. In patients with inflammatory diseases, 64Cu-DOTA-ECL1i PET revealed specific detection of CCR2+ cells in inflammatory tissues. In a rat AAA model, 64Cu-DOTA-ECL1i PET revealed specific localization within the aneurysm, as well as sensitive detection of CCR2+ inflammatory cells. Human AAA specimens demonstrated specific binding of 64Cu-DOTA-ECL1i to CCR2 by autoradiography. Thus, we hypothesize that 64Cu-DOTA-ECL1i detect CCR2+ cells mediated aneurysmal activity and can be utilized for AAA molecular imaging. We propose to assess the potential of 64Cu-DOTA-ECL1i as a biomarker for AAA patients imaging.

ELIGIBILITY:
Inclusion Criteria:

* 40 years old and above
* With or without active tobacco use
* Asymptomatic patients with known AAAs by CT angiogram (men ≥ 5.5 cm, women ≥ 5.0cm).
* Non-AAA volunteers will have a documented absence of AAA by exam and recent screening ultrasound (US).
* Able to comprehend and willing to follow instructions for the study procedures as called for by the protocol

Exclusion Criteria:

* Inability to receive and sign informed consent.
* Patients with Stage ≥ 4 chronic renal failure (calculated by modification of diet in renal disease eGFR equation [to minimize confounding imaging variables])
* Documented allergy to iodinated contrast and/or shellfish.
* Patients with an unstable clinical condition that in the opinion of the principal investigators or designee precludes participation in the study.
* Inability to tolerate 60 minutes in a supine position with arms down at sides, as necessary for PET/CT.
* Positive pregnancy test or lactating.
* Other conditions such as symptomatic/recently treated coronary disease, cancer requiring oncologic management, or autoimmune/inflammatory diseases (e.g., rheumatoid arthritis or multiple sclerosis) that are known to have increased associated CCR2 expression.
* Non-AAA volunteers may not carry a diagnosis of aortoiliac occlusive disease, as documented by their treating vascular surgeon, as significantly progressed atherosclerotic disease may demonstrate exaggerated, associated CCR2 expression.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Determine the binding characteristics of 64Cu-DOTA-ECL1i in ex vivo human AAA specimens and correlate with associated histopathological features | 4 years
  Perform histopathological evaluation of human AAA specimens and categorize them based on clinical status (e.g, diameter) and degree of inflammation. The investigators will consider healthy, nonatherosclerotic aorta as negative controls, and non-aneurysmal aortas from patients that have undergone surgery for aortoiliac occlusive disease as positive controls. Disease severity will be graded as mild, moderate, and severe based on the degree of VSMC loss and elastic layer disruption (<25%, 25-75%, and >75% compared to normal aorta). The presence of atherosclerotic changes, intraluminal thrombus and degree and location of associated inflammation will be documented.
  The degree of inflammation will be scored in three tiers: absent/minimal (rare scattered inflammatory cecells), moderate (small clusters of inflammatory cells), and severe (easily identified with scanning magnification).
Determine the relationship between 64Cu-DOTA-ECL1i binding, regional CCR2 gene expression, cytokine profiles and local matrix metalloproteinase (MMP) activity. | 4 years
  Tissue will be collected from patients who undergo surgery and tissue will be collected from a repository at our institution. Investigators will correlate level of MMP expression, activity and cytokine profiles of each specimen, with associated histopathological features. To address the concern of tissue heterogeneity, investigators will perform spatial transcriptomics assays for quantitative measurement of regional CCR2 gene expression on human AAA sections. Since clinical status and aneurysmal anatomic features on preop imaging of each patient is known, investigators will explore correlation of standard of care imaging findings with those from Aim 2A and this sub-aim to determine the role of CCR2 in AAA pathogenesis and its potential as a biomarker for human AAA disease.
Assess the 64Cu-DOTA-ECL1i imaging characteristics in AAA patients undergoing open repair and non-AAA volunteers to determine the relationship between tracer uptake and molecular characterization of prospectively collected AAA tissues. | 4 years
  Investigators will determine retention of 64Cu-DOTA-ECL1i in abdominal aorta of non-AAA volunteers (n=10, 5 women and 5 men). Investigators will image AAA patients pre-operatively and collect tissue at the time of open repair in an attempt to demonstrate ex-vivo tissue corroboration of our imaging findings (n=20, 10 women and 10 men).
Assess imaging reproducibility of 64Cu-DOTA-ECL1i PET/CT in non-surgical AAA patients. | 4 years
  Reproducibility group - Aim 3B, We will demonstrate consistent 64Cu-DOTAECL1i uptake by performing repeated imaging studies in a separate group of non-surgical AAA patients (n=20, 10 women and 10 men). Completion of this sub-aim will provide support for the use of 64Cu-DOTA-ECL1i PET for evaluating AAA disease in a reliable fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M. Zayed, MD, Principal Investigator — Washington University of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT04586452/ICF_000.pdf